CLINICAL TRIAL: NCT02386592
Title: Prevention of Nosocomial Bacteremia and Mortality Among Neonates at a Tertiary Referral Center in Zambia
Brief Title: Prevention of Nosocomial Bacteremia Among Zambian Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); Zambia Center for Applied Health Research and Development (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-33473
Record Dates: First submitted 2015-02-17; First posted 2015-03-12 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Neonatal Sepsis; Neonatal Mortality
MeSH Terms: conditions — Neonatal Sepsis | interventions — chlorhexidine gluconate; Hand Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Infection control package consisting of alcohol hand rub hand hygiene (HH), 2% chlorhexidine gluconate (CHG) body washes, infection control training, and text messages with basic Infection control reminders via SMS text
  Interventions: Drug: Chlorhexidine gluconate (CHG); Behavioral: Hand hygiene (HH); Behavioral: Infection control training; Other: Infection control reminders via SMS text

INTERVENTIONS:
Drug: Chlorhexidine gluconate (CHG) — All enrolled neonates admitted to the NICU during the implementation and intervention periods will undergo CHG bathing (sparing head and face) at the time of admission at and thereafter once weekly.
  Other Names: 2% chlohexidine gluconate body wash
Behavioral: Hand hygiene (HH) — Alcohol hand rub will be produced in the hospital pharmacy and will be readily available in the NICU (via wall-mounted dispensers) throughout the intervention period. Hand hygiene among NICU physicians and nurses will actively be promoted through the intervention period.
Behavioral: Infection control training — All NICU healthcare workers will receive infection prevention training which will involve structure training on HH, universal precautions, neonatal skin antisepsis and peripheral IV placement and line care.
Other: Infection control reminders via SMS text — Infection control practice reminders will be sent to NICU healthcare workers on a daily basis via SMS messages.

SUMMARY:
The purpose of this study is to estimate the burden of disease, identify risk factors associated with nosocomial bacteremia among neonates and assess the efficacy of low-cost measures targeted to known and suspected nosocomial BSI (bloodstream) risk factors, the investigators propose to study the impact of a novel package of infection control interventions on nosocomial bacteremia and mortality among neonates at a tertiary care center in sub-Saharan Africa.

DETAILED DESCRIPTION:
The study is an18 month prospective quasi-experimental evaluation of nosocomial bacteremia and mortality among hospitalized neonates and will consist of a 6-month baseline period to capture the incidence and all-cause mortality of nosocomial BSIs, a 1-month implementation period of low-cost infection control strategies (including alcohol-based hand rub [AHR], 2% chlorhexidine gluconate [CHG], hospital staff education and text message-based reminders of infection control recommendation) and an 11-month intervention period.

All neonates admitted to the neonatal intensive care unit (NICU) of the University Teaching Hospital (UTH) in Lusaka, Zambia during the study period will be eligible for study enrollment. This study will determine the capacity of an innovative bundle of low cost, simple and locally available interventions that leverage new technologies and expand application of highly effective interventions in order to reduce the incidence of nosocomial bacteremia among NICU patients in a developing country setting.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the study site NICU during the study period (including both "inborn" and "outborn" neonates)

Exclusion Criteria:

* Neonates without documented birth date
* Parent or guardian unavailable or unwilling to provide consent

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9410 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
All-cause neonatal mortality in hospitalized neonates | 18 months
  in hospitalized neonates at University Teaching Hospital (UTH), a large tertiary referral center, in Zambia before and after the introduction of low-cost infection-control interventions.

SECONDARY OUTCOMES:
Incidence of nosocomial bacteremia in hospitalized neonates | 18 months
  Incidence of nosocomial bacteremia in hospitalized neonates at UTH before and after the introduction of low-cost infection-control interventions.
Attributable risk of maternal, neonatal, hospital factors and nosocomial bacteremia among hospitalized neonates | 18 months
  Measure the attributable risk of maternal, neonatal and hospital factors as well as invasive procedures on nosocomial bacteremia among neonates hospitalizedat UTH
Prevalence of nosocomial bacteremia caused by MDR-GNR infections among hospitalized neonates | 18 months
  Prevalence of nosocomial bacteremia caused by MDR-GNR infections among neonates at UTH.

CONTACTS AND LOCATIONS:
Overall Officials: Davidson H Hamer, MD, Principal Investigator — BU School of Medicine
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
We are willing to share participant and microbiological data after publication of the main study findings and after receipt of an acceptable analysis plan.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after publication of the main study findings and full microbiological analysis
Access Criteria: Upon receipt and review of an acceptable proposal for analysis of the data, we will share the database.

REFERENCES:
- [Background] Gill CJ, Mantaring JB, Macleod WB, Mendoza M, Mendoza S, Huskins WC, Goldmann DA, Hamer DH. Impact of enhanced infection control at 2 neonatal intensive care units in the Philippines. Clin Infect Dis. 2009 Jan 1;48(1):13-21. doi: 10.1086/594120. PMID 19025496
- [Background] Aiken AM, Mturi N, Njuguna P, Mohammed S, Berkley JA, Mwangi I, Mwarumba S, Kitsao BS, Lowe BS, Morpeth SC, Hall AJ, Khandawalla I, Scott JAG; Kilifi Bacteraemia Surveillance Group. Risk and causes of paediatric hospital-acquired bacteraemia in Kilifi District Hospital, Kenya: a prospective cohort study. Lancet. 2011 Dec 10;378(9808):2021-2027. doi: 10.1016/S0140-6736(11)61622-X. Epub 2011 Nov 29. PMID 22133536
- [Background] Milstone AM, Elward A, Song X, Zerr DM, Orscheln R, Speck K, Obeng D, Reich NG, Coffin SE, Perl TM; Pediatric SCRUB Trial Study Group. Daily chlorhexidine bathing to reduce bacteraemia in critically ill children: a multicentre, cluster-randomised, crossover trial. Lancet. 2013 Mar 30;381(9872):1099-106. doi: 10.1016/S0140-6736(12)61687-0. Epub 2013 Jan 28. PMID 23363666
- [Derived] Mwananyanda L, Pierre C, Mwansa J, Cowden C, Localio AR, Kapasa ML, Machona S, Musyani CL, Chilufya MM, Munanjala G, Lyondo A, Bates MA, Coffin SE, Hamer DH. Preventing Bloodstream Infections and Death in Zambian Neonates: Impact of a Low-cost Infection Control Bundle. Clin Infect Dis. 2019 Sep 27;69(8):1360-1367. doi: 10.1093/cid/ciy1114. PMID 30596901